CLINICAL TRIAL: NCT04268017
Title: Reliability and Competing Validity of the FeetMe Monitordevice® Measurement of the Spatial-temporal Parameters of the gaitRite System® in Healthy Subjects
Brief Title: Validation Study : FeetMe® Monitor Insoles for the Evaluation of Gait Speed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FeetMe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FTM_HEALTHY_01
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Gait analysis; FeetMe®; GaitRite®; Healthy; Validation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Experimental)
  Interventions: Device: FeetMe Monitor

INTERVENTIONS:
Device: FeetMe Monitor — For gait parameters' evaluation, the investigator asks the participant to move in a straight line over a 10-meter mat. The participant had to start the feet in line and then start walking at a comfortable speed. During this time, the investigator records the gait parameters from the FeetMe Monitor® and Gaitrite® system.
  An operator asked the patient to repeat 3 trials. The same sequence was repeated by three other operators. The same measurement is done 7 days later.
  A questionnaire is given to assess the ergonomics of the device

SUMMARY:
The aim of this study is to validate a smart insoles system in comparison to the gold-standard GaitRite in a healthy population. The device evaluate gait parameters in real time thanks to an embedded algorithm based on the processing of inertial measurement unit and 19 sensors signals.

At D0 and D7, the volunteer is evaluated by both the GaitRite® system and the FeetMe Monitor® system simultaneously. Healthy volunteers have two measurements 7 days apart. The volunteer repeats 5 trials at a comfortable speed on the GaitRite® mat while wearing the FeetMe® insoles. Each measurement is repeated by 4 different operators. A total of 20 trials are made by the volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Have more than 18 years old
* Don't be pregnant or breast feeding

Exclusion Criteria:

* Be part of another study
* Not be able to give consent
* Not have access to social security

Min Age: 18 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Velocity measured through FeetMe Monitor device and GaitRit | 1 day

SECONDARY OUTCOMES:
Stride length measured through FeetMe Monitor device and GaitRite | 1 day
Cadence measured through FeetMe Monitor device and GaitRite | 1 day
Stance phase measured through FeetMe Monitor device and GaitRite | 1 day
Swing phase measured through FeetMe Monitor device and GaitRite | 1 day
Stride duration measured through FeetMe Monitor device and GaitRite | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Fédération de Rééducation Neurolocomotrice, Laboratoire ARM - Hôpital Henri MONDOR, Assistance Publique - Hôpitaux de Paris, Créteil, France

IPD SHARING:
Plan to Share IPD: No